CLINICAL TRIAL: NCT02399436
Title: Appalachians Together Restoring the Eating Environment
Acronym: Appal-TREE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark Swanson, PhD (Other)
Collaborators: Community Farm Alliance (Other)
Responsible Party: Sponsor-Investigator, Mark Swanson, PhD, Associate Professor, Department of Health Behavior, College of Public Health, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12-0900-P3H
Record Dates: First submitted 2015-03-12; First posted 2015-03-26 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Dietary Habits
Keywords: Community-Based Participatory Research; Community-Institutional Relations
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- School-Based Healthy Snacking Campaign (Experimental): Students who attend middle and high schools in the experimental county that participate in the healthy snacking campaign intervention.
  Interventions: Behavioral: School-Based Healthy Snacking Campaign
- Comparison Schools (No Intervention): Students who attend middle and high schools in the comparison county, which does not receive any intervention components.
- Community Cooking Classes (Experimental): Adults in the intervention county who enroll in group cooking classes (single-group pretest-posttest)
  Interventions: Behavioral: Community Cooking Classes

INTERVENTIONS:
Behavioral: School-Based Healthy Snacking Campaign — The school-based healthy snacking campaign includes the following activities:
  * Sales promotion of snack choices that meet federal Smart Snack guidelines during the school day and at school events, such as snack bars and after-school events;
  * The installation of new filtered water fountains outfitted with water-filling stations;
  * The distribution of re-usable water bottles to students at participating schools; and
  * A social marketing campaign to support adoption of the healthy snacks and water consumption by students.
  Arms: School-Based Healthy Snacking Campaign
Behavioral: Community Cooking Classes — Cooking classes will be delivered to groups of 8-12 adult participants as a series of 8 weekly classes in community venues. The content of each class is driven by topics and themes identified and prioritized by community members, namely cooking healthy on tight budget.
  Arms: Community Cooking Classes

SUMMARY:
Most of the nation's serious chronic health challenges and causes of death, including diabetes, heart disease, cancer, and obesity, are directly linked to sub-optimal diet. Both poor diets and associated disease are disproportionately common in the Appalachian counties of eastern Kentucky, a region with stark health inequities, including elevated rates of obesity, overweight, and premature mortality. The purpose of this pilot study is to evaluate a multi-component intervention developed through community-based participatory research methods for improving access to healthy foods and enhancing dietary intake in eastern Kentucky. The intervention components evaluated in this study consist of a social marketing campaign delivered to middle and high schools to promote healthy snacking and water consumption, and a series of group cooking classes for adults.

DETAILED DESCRIPTION:
This pilot study evaluates two principal components of a community-based intervention to improve dietary habits and access to healthy foods: a school-based healthy snacking campaign and a series of community cooking classes for adults. The primary outcome assessed within each intervention component is dietary intake as measured by self-reported beverage and food consumption in pre-post surveys. Secondary outcome variables include attitudes, preferences, confidence, self-efficacy and other psychosocial variables related to healthy eating behaviors, perceptions of healthy food availability, food purchasing and preparation habits, and perceived barriers to healthy eating.

The school-based intervention component employs a nonequivalent control group research design. A subset of middle- and high-schools within a single county in eastern KY will receive a healthy snacking campaign intervention, and students from randomly selected classrooms within these schools will be invited to enroll in the study. Students from middle- and high-school classrooms in a comparison county that receives no intervention will serve as nonequivalent controls. The investigators specific aims for this component are to improve the availability of healthy snack foods that students may purchase at school, increase student consumption of healthy snacks over unhealthy snacks, and increase the consumption of water over sugar-sweetened beverages. Following baseline, posttest surveys will be administered at 3, 6 and 14 months.

Community cooking classes will be delivered to a non-random sample of adults who will complete pretest-posttest measures at baseline and 8 weeks. The specific aims of this component are to increase the consumption of healthy foods at home, and increase participant knowledge, skills, and self-efficacy around healthy home cooking.

ELIGIBILITY:
Inclusion Criteria:

* For School-Based Component: 6th-12th grade students enrolled in a participating school and classroom in the intervention or comparison county.
* For Cooking Classes: Adults aged 18 years and older residing in intervention county who have at least one juvenile in household.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Beverage Consumption (Students) | Baseline, 3 months, 6 months, and 14 months
  Frequency and quantity of beverages consumed in past month. Includes water, 100% fruit juice, sugar-sweetened beverages, sugar-free beverages and milk.
Change in Snack Consumption (Students) | Baseline, 3 months, 6 months, and 14 months
  Frequency and quantity of snacks consumed in past month. Includes chips (regular and low-fat), salty snacks, candy, desserts, vegetables, fruit, nuts and seeds, vegetable dips, yogurt, and popcorn.
Change in Dietary intake (Adults) | Baseline to 8 weeks
  Frequency of consumption of fruits, vegetables, beans, candy, pastries, desserts, and salty snacks in the past month.

SECONDARY OUTCOMES:
Change in Snacking Attitudes and Preferences (Students) | Baseline, 3 months, 6 months, and 14 months
  Survey items address taste preferences, attitudes about healthy eating behaviors and body image
Change in Healthy Snacking Confidence and Self-efficacy (Students) | Baseline, 3 months, 6 months, and 14 months
Change in Availability of Healthy Snack Foods (Students) | Baseline, 3 months, 6 months, and 14 months
  Frequency of availability of healthy and unhealthy snack foods at school
Change in Snack Food Purchasing Habits (Students) | Baseline, 3 months, 6 months, and 14 months
  Frequency of purchasing snack foods and beverages at fast food restaurants, convenience stores, and school venues and events
Change in Food Preparation Habits (Adults) | Baseline to 8 weeks
  Likelihood of performing healthy food preparation behaviors; survey items address meal planning and preparation
Change in Food Purchasing Habits (Adults) | Baseline to 8 weeks
  Frequency of purchasing food at work, grocery/convenience stores, restaurants and produce stands
Change in Perceptions of Availability of Healthy Foods (Adults) | Baseline to 8 weeks
  Survey items address availability of high quality fruits and vegetables and low-fat foods
Change in Barriers to Healthy Eating (Adults) | Baseline to 8 weeks
  Survey items address physical, psychosocial, emotional, and financial barriers to healthy eating

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States